CLINICAL TRIAL: NCT06295211
Title: Brentuximab Vedotin Combined With Bendamustine Supercharge, a Low-toxicity and Efficient Salvage Regimen for Primary Refractory or First-relapsed Classic Hodgkin Lymphoma: Long-term Results of a Retrospective Monocenter Study.
Acronym: HL_PR/R-B
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Marco Picardi, professor, Federico II University
Other Study IDs: FEDII_HL_PR/R-Bv-Bs
Record Dates: First submitted 2024-02-23; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Hodgkin Lymphoma
Keywords: Hodgkin lymphoma; primary refractory; bendamustine supercharge; brentuximab vedotin
MeSH Terms: conditions — Hodgkin Disease | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational — observational

SUMMARY:
This is a retrospective, monocenter and non-interventional study. Data were retrospectively collected from all patients who completed the BV-Bs scheme in the time period between 1 September 2013 and 1 September 2023.

DETAILED DESCRIPTION:
This is a retrospective, monocenter and non-interventional study. Data were retrospectively collected from all patients who completed the BV-Bs scheme in the time period between 1 September 2013 and 1 September 2023.

The regimen consisted of 3-day outpatient intravenous infusions of 1.8 mg/kg Bv on Day 1 of each 3-week cycle (as established by Younes and colleagues) sequentially combined with bendamustine (at least 24 hours after Bv, precisely on days 2 and 3 of the treatment cycle; as reported by Picardi et al) at a fixed dose of 120 mg/m2 per day.

All patients who achieved at least partial remission were considered eligible for peripheral blood stem cell (PBSC) collection (performed with granulocyte colony-stimulating factor [G-CSF] and endoxan or plerixafor, if necessary) and proceeded to ASCT at any time beyond cycle 4.

The anti-tumor activity of this treatment regimen was assessed according to the Lugano criteria at the end of the combination treatment.

Prior to the first cycle of Bv-Bs, all patients underwent a clinical evaluation that included assessment of B symptoms, World Health Organization performance status, and measurement of palpable lesions. In particular, imaging procedures were conducted after the second and fourth cycles or prior to ASCT. The response was based on international criteria (Cheson et al, 2016). PET scans were considered positive or negative based on the Deauville 5-point scale criteria.

ELIGIBILITY:
Inclusion Criteria:

* patients age between 18 years and 60 years;
* histological confirmation of CD30+ subtype cHL at first relapse or at refractory (patients who have failed to achieve complete remission at the end of treatment with 4-6 cycles of ABVD or who have progressed early during front-line treatment [after 2 cycles of ABVD] with interim FDG-PET/CT with Deauville scale score of 5 [primary refractory patients])
* treatment with at least 1 cycle of Bs and Bv at doses of 120 mg/m2 and 1.8 mg/kg, respectively
* metabolically active disease measurable at fluoro-desossi-glucose-positron emission tomography/computed tomography (FDG-PET/CT)
* EGOG performance status 0-2 (or 3, if due to illness).

Exclusion Criteria:

* patients not fulfilling inclusion criteria

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This is a retrospective, monocenter and non-interventional study. Data were retrospectively collected from all patients who completed the BV-Bs scheme in the time period between 1 September 2013 and 1 September 2023.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Overall survival | 10 year period
  survival

SECONDARY OUTCOMES:
Progression overall survival | 10 year period
  survival
Response to treatment | at end of 4 cycles treatment (each cycle of 28 days)
  Complete Metabolic Remission rate
Incidence of treatment emergent adverse events | during 4 cycles of treatment (each cycle of 28 days)
  side effect to regimen related to both Brentuximab and bendamustine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Picardi M, Della Pepa R, Giordano C, Pugliese N, Mortaruolo C, Trastulli F, Rascato MG, Cappuccio I, Raimondo M, Memoli M, Monteverde M, Mascolo M, Pane F. Brentuximab vedotin followed by bendamustine supercharge for refractory or relapsed Hodgkin lymphoma. Blood Adv. 2019 May 14;3(9):1546-1552. doi: 10.1182/bloodadvances.2019000123. PMID 31088808
- [Result] Cheson BD, Ansell S, Schwartz L, Gordon LI, Advani R, Jacene HA, Hoos A, Barrington SF, Armand P. Refinement of the Lugano Classification lymphoma response criteria in the era of immunomodulatory therapy. Blood. 2016 Nov 24;128(21):2489-2496. doi: 10.1182/blood-2016-05-718528. Epub 2016 Aug 29. PMID 27574190